CLINICAL TRIAL: NCT02117453
Title: Multicenter, Prospective, Randomized, Controlled, Double-blind Trial on the Impact of Rosuvastatin on Subclinical Markers of Atherosclerosis in Patients With Primary Necrotizing Vasculitides
Acronym: STATVAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P120127; 2013-002531-15 (EudraCT Number)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: ANCA-associated Primary Necrotizing Vasculitides
Keywords: ANCA vasculitis; Statin; Subclinical markers of atherosclerosis; Cardiovascular events; Myocardial infarction; Stroke; Arterial revascularization; Unstable angina; Death
MeSH Terms: conditions — Myocardial Infarction; Stroke; Angina, Unstable; Death | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): Rosuvastatin 20 mg/day
  Interventions: Drug: Rosuvastatin
- Group II (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20 mg/day
  Arms: Group I
Drug: Placebo — Placebo
  Arms: Group II

SUMMARY:
The purpose of this study is to assess whether rosuvastatin could reduce the subclinical markers of atherosclerosis and the incidence of major cardiovascular events in patients with primary necrotizing vasculitides.

DETAILED DESCRIPTION:
Previous studies demonstrated the presence of subclinical atherosclerosis in patients with ANCA-associated systemic necrotizing vasculitis. Since statins lower levels of inflammatory proteins and cholesterol, we hypothesized that people with ANCA-associated systemic necrotizing vasculitis but without indication for statin treatment according to recommandations might benefit from statin treatment.

ELIGIBILITY:
Inclusion Criteria:

Patient > 18 years. ANCA-associated vasculitis: granulomatosis with polyangiitis (GPA), microscopic polyangiitis (MPA) and eosinophilic granulomatosis with polyangiitis (EGPA, Churg-Strauss syndrome).

Patients will fulfill the Chapel Hill Consensus Criteria and the American College of Rheumatology criteria, in remission of vasculitis.

Patients in remission of vasculitis after induction therapy (for first flare or relapse), including corticosteroids associated or not with immunosuppressive agents according to Good Clinical Practice for the treatment of vasculitis, between 6 months and 10 years after the beginning of induction therapy.

Patients with informed and signed consent

Exclusion Criteria:

Other systemic vasculitis. Secondary vasculitis (paraneoplastic or infectious). Patient with active vasculitis after induction therapy, requiring salvage therapy.

Inability to sign informed consent. Inability to take the experimental treatment. Hypersensitivity to rosuvastatin or to any of the excipients. Pregnancy. Chronic HCV, HBV and/or HIV infection. Patient receiving other statin or other hypolipemic agent. Patient requiring treatment with statin according to Afssaps recommandations published in 2005 as primary or secondary prevention.

Subclinical atherosclerosis that confers a high cardiovascular risk before patient randomization :

* Carotid stenosis greater than 50% in diameter
* Ectasia of the abdominal aorta
* Intima-media thickening greater than 1.2 mm
* Diffuse atherosclerosis lesions
* Heterogeneous or hypoechoic prominent plaques greater than 2 mm

Participation in another interventional study within 3 months before inclusion. Sick patients will not be excluded if they participate simultaneously in a strictlu observational study or a study with only blood samplings.

Any medical or psycatric disease that could prevent from administrating drugs or from following-up the patient according to the protocol, and/or that would expose the patient to an important number of side effects, according to the principal investigator.

Non affiliation to a social security system or any social protection system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in mean carotid intima-media thickness for 2 predefined sites (distal common carotid arteries) | 24 months
  Assessed with B-mode ultrasound

SECONDARY OUTCOMES:
Annualized rate of change in mean carotid intima-media thickness for 2 predefined sites (distal common carotid arteries) | 24 months
  Assessed with B-mode ultrasound
Mean change from baseline in the number of plaques in three peripheral vessels (carotid and femoral arteries and abdominal aorta) at 6, 12 and 24 months | 24 months
  Assessed with B-mode ultrasound
Mean change from baseline in serum biomarkers of subclinical atherosclerosis at 6, 12 and 24 months | 24 months
  ultra-sensitive CRP, VCAM-1, P-selectin, thrombomodulin
Rate of major cardiovascular events (myocardial infarction, stroke, arterial revascularization, hospitalization for unstable angina, or death from cardiovascular causes) | 24 months
Rate of vasculitis relapses defined by BVAS>0 | 24 months
Rate of adverse events | 24 months
Mean change from baseline in lipid profile (triglycerids, total, HDL and LDL cholesterol) at 6, 12 and 24 months compared to baseline value. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Terrier, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Loic Guillevin, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No